CLINICAL TRIAL: NCT02683616
Title: Fatty Acid Metabolism in Obstructive Sleep Apnea (FAMOSA)
Acronym: FAMOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Jan Polak, Associate Professor, Faculty Hospital Kralovske Vinohrady
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZV15_30155A
Record Dates: First submitted 2016-02-09; First posted 2016-02-17 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Sleep Apnea; Fatty Acid Metabolism; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- OSA + T2DM (Experimental): CPAP treatment
  Interventions: Device: CPAP
- OSA no T2DM (Experimental): CPAP treatment
  Interventions: Device: CPAP
- T2DM no OSA (No Intervention): Standard care
- Healthy controls no ÓSA (No Intervention): no intervention

INTERVENTIONS:
Device: CPAP — Continuous Positive Airway Pressure in cases of moderate/severe OSA
  Arms: OSA + T2DM; OSA no T2DM

SUMMARY:
Obstructive sleep apnea syndrome (OSA) is a disease affecting 5-15% of population and 50-80% of type 2 diabetes mellitus (T2DM) and obese subjects. OSA causally contributes to the development of glucose intolerance and T2DM. The project is targeting the gap in providing effective treatment of metabolic impairments associated with OSA, particularly T2DM. In contrast to proved benefits of OSA treatment with CPAP (continuous positive airway pressure) on cardiovascular morbidity/mortality, studies on the impact of CPAP on diabetes control are disappointing. In fact, OSA-induced metabolic impairments might not be reversible with CPAP treatment, as investigators suggested recently. Clearly, the search for additional treatments, probably pharmacological, is warranted. Investigators hypothesize that elevated levels of free fatty acids (FFA), as detected in OSA patients, are linking OSA with the T2DM development. The aim of the study is to target adipose tissue and muscle dysfunction leading to elevated FFA and develop thus novel pharmacological treatments based on lipolysis inhibition and stimulation of FFA oxidation.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus
* Age 18 - 85 years
* BMI 22-40 kg/m2
* moderate or severe OSA diagnosed by home sleep study

Exclusion Criteria:

* treatment with insulin
* other acute or chronic endocrine or inflammatory disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Glycerol release (lipolysis) in adipose tissue | Baseline and 6 months
  Changes in interstitial glycerol concentration in adipose tissue
Palmitate oxidation in skeletal muscle | Baseline and 6 months
  Changes in palmitate oxidation in muscle biopsies measured ex vivo

CONTACTS AND LOCATIONS:
Locations (1):
- FN Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No